CLINICAL TRIAL: NCT06707818
Title: Psychosocial Factors and Postoperative Pain in Aesthetic Breast Surgery: A Prospective Observational Study
Brief Title: Psychosocial Factors and Postoperative Pain in Aesthetic Breast Surgery
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Murat Tümer, MD, Anesthesiologist, V.K.V. American Hospital, Istanbul
Other Study IDs: PostopPainAndPsychology
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Psychological Factors; Breast Surgery; Aesthetic Surgery; Anesthesia, General; Quality of Recovery (QoR-15); Patient Satisfaction; Pain Management
Keywords: Postoperative pain; Aesthetic breast surgery; psychosocial factors; pain management
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for aesthetic breast surgery: This group includes patients undergoing aesthetic breast surgery between January 2024 and January 2025 who are assessed preoperatively, intraoperatively, and postoperatively.
  Interventions: Other: Preoperative Interventions; Other: Intraoperative Interventions; Other: Postoperative Interventions

INTERVENTIONS:
Other: Preoperative Interventions — During the initial surgical consultation, participants will provide informed consent. Demographic data and several validated assessment scales will be collected, including the Perceived Socioeconomic Status Scale (8), Ten-Item Personality Inventory (9), Pain Catastrophizing Scale (10), Hospital Anxiety and Depression Scale (11), Rosenberg Self-Esteem Scale (12), Quality of Recovery-15 (QoR-15) questionnaire (13), and the Visual Analog Scale (VAS) for pain (14).
Other: Intraoperative Interventions — All surgical procedures will follow the standard general anesthesia protocol of the hospital. General anesthesia induction will involve propofol (1-2 mg/kg), fentanyl (1 mcg/kg), and rocuronium (0.6 mg/kg) for endotracheal intubation. Anesthesia maintenance will be performed with desflurane (4-6%) and remifentanil (0.1 mcg/kg/min), with adjustments as needed based on blood pressure and heart rate. Post-induction, dexamethasone (4 mg) will be administered for anti-inflammatory effects. To support postoperative pain management, tramadol (1 mg/kg), ibuprofen (400 mg), and paracetamol (1 g) will be administered before the end of the procedure. Ondansetron (4 mg) will be used for nausea prophylaxis. All intraoperative medications and dosages will be recorded without intervention.
Other: Postoperative Interventions — In the recovery room, analgesic interventions will follow the hospital's standard protocol: patients with VAS scores between 3 and 7 will receive 25 mcg of fentanyl, while those with scores above 7 will receive 50 mcg.
  All patients will receive standard multimodal analgesia during the ward stay, including paracetamol (1 g, three times daily) and ibuprofen (400 mg, twice daily). Patient-controlled analgesia (PCA) devices will administer tramadol (10 mg IV per patient request, without continuous infusion).

SUMMARY:
This study investigates the relationship between psychosocial factors, particularly self-esteem and personality traits, and postoperative pain in patients undergoing aesthetic breast surgery. Previous research suggests that psychological factors like depression, anxiety, and low self-esteem may influence pain perception. The study aims to contribute to personalized pain management strategies for these patients.

A prospective, observational cohort study will be conducted at VKV American Hospital from January 2024 to January 2025. Eligible participants (18+ years old, ASA status 1-3) will be assessed preoperatively using validated scales for self-esteem, personality traits, anxiety, depression, and pain perception. Intraoperative procedures will follow a standardized anesthesia protocol, with pain and recovery data collected postoperatively. Pain scores and medication usage will be recorded, and patient satisfaction will be assessed using the Quality of Recovery-15 scale.

This study seeks to enhance understanding of psychological influences on postoperative pain, potentially improving pain management protocols for aesthetic surgery patients.

DETAILED DESCRIPTION:
INTRODUCTION Pain is an unpleasant experience associated with actual or potential tissue damage, involving sensory, emotional, cognitive, and social components (1). There are studies in the literature that examine the relationship between postoperative acute pain and psychological factors (2, 3). For example, studies in cancer patients undergoing reconstructive breast surgery have shown that depression, anxiety levels, and abnormal pain perception (pain catastrophizing) are associated with postoperative pain (4). Psychological factors that could influence pain in aesthetic surgeries may be more diverse. Self-esteem and personality types are among the psychological factors that could affect pain.

Self-esteem refers to an individual's beliefs and perceptions about themselves. It plays a significant role in shaping an individual's thoughts about their physical appearance. People with low self-esteem are generally dissatisfied with their appearance, which may lead them to seek aesthetic surgery as a way to improve their self-worth. Low self-esteem has been associated with an increased likelihood of undergoing aesthetic surgery (5). Furthermore, aesthetic surgeries have been linked to significant improvements in self-esteem. A systematic review conducted by Javo and colleagues (2019) showed that more than 70% of aesthetic surgery patients experienced significant increases in self-esteem (6).

Another factor that could be related to pain is personality traits. Studies have shown that personality traits are important predictors of postoperative pain and complications in aesthetic surgeries (7). Traits such as perfectionism, neuroticism, and anxiety have been associated with increased postoperative pain and poor surgical outcomes. Individuals with these traits may experience anxiety and fear before surgery, leading to a lower pain threshold and increased sensitivity to pain sensations.

Aesthetic surgery is a rapidly growing industry worldwide. The desire for physical recovery and maintaining a youthful appearance has led to an increase in demand for aesthetic surgeries. However, the psychological effects of these surgeries and their relationship with pain have not been fully investigated. The aim of our study is to examine the relationship between psychosocial factors, particularly self-esteem and personality types, and postoperative pain in patients undergoing aesthetic breast surgery. This study is expected to contribute to the literature on developing personalized pain management strategies for aesthetic surgery patients.

To investigate the relationship between self-esteem, personality types, other psychosocial factors, and postoperative pain in patients undergoing aesthetic breast surgery. To contribute to the literature on the development of personalized pain protocols for aesthetic surgery patients.

METHOD After obtaining ethical approval from the Koç University Committee on Human Research, with approval number [2023.305.IRB1.101], a prospective, observational cohort study will be conducted at VKV American Hospital. Patients scheduled for aesthetic breast surgery between January 2024 and January 2025 will be informed about the study and invited to participate. Participants eligible for inclusion in the study must be aged 18 years or older and have an American Society of Anesthesiologists (ASA) physical status classification of 1-3. Individuals will be excluded if they are under the age of 18, have an ASA status of 4, decline to participate, or have a history of anxiety disorders and/or psychological conditions.

The study will include three main phases: preoperative, intraoperative, and postoperative periods. The data collected from these periods will be used to evaluate perioperative outcomes, including pain management efficacy, recovery quality, and overall patient satisfaction.

1. Preoperative Period:

   One week before surgery, during the initial surgical consultation, participants will provide informed consent. Demographic data and several validated assessment scales will be collected, including the Perceived Socioeconomic Status Scale (8), Ten-Item Personality Inventory (9), Pain Catastrophizing Scale (10), Hospital Anxiety and Depression Scale (11), Rosenberg Self-Esteem Scale (12), Quality of Recovery-15 (QoR-15) questionnaire (13), and the Visual Analog Scale (VAS) for pain (14).
2. Intraoperative Period:

   All surgical procedures will follow the standard general anesthesia protocol of the hospital. General anesthesia induction will involve propofol (1-2 mg/kg), fentanyl (1 mcg/kg), and rocuronium (0.6 mg/kg) for endotracheal intubation. Anesthesia maintenance will be performed with desflurane (4-6%) and remifentanil (0.1 mcg/kg/min), with adjustments as needed based on blood pressure and heart rate. Post-induction, dexamethasone (4 mg) will be administered for anti-inflammatory effects. To support postoperative pain management, tramadol (1 mg/kg), ibuprofen (400 mg), and paracetamol (1 g) will be administered before the end of the procedure. Ondansetron (4 mg) will be used for nausea prophylaxis. All intraoperative medications and dosages will be recorded without intervention.
3. Postoperative Period:

In the recovery room, pain scores will be recorded at 0, 30, and 60 minutes postoperatively by blinded nurses. Analgesic interventions will follow the hospital's standard protocol: patients with VAS scores between 3 and 7 will receive 25 mcg of fentanyl, while those with scores above 7 will receive 50 mcg. The total fentanyl dosage and any side effects, such as nausea, respiratory difficulty, or shivering, will be documented.

All patients will receive standard multimodal analgesia during the ward stay, including paracetamol (1 g, three times daily) and ibuprofen (400 mg, twice daily). Patient-controlled analgesia (PCA) devices will administer tramadol (10 mg IV per patient request, without continuous infusion). Data on VAS scores at 6 and 24 hours postoperatively, as well as the total tramadol dosage administered via PCA, will be recorded. Additionally, participants' satisfaction with pain management will be assessed using the Quality of Recovery-15 scale at 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have an American Society of Anesthesiologists (ASA) physical status classification of 1-3.

Exclusion Criteria:

* under the age of 18,
* have an ASA status of 4,
* history of anxiety disorders and/or psychological conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for aesthetic breast surgery between January 2024 and January 2025 will be informed about the study and invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Preoperatively and 24 hours postoperatively.
  Participants' satisfaction with pain management will be assessed using the Quality of Recovery-15 scale preoperatively and 24 hours postoperatively.
  The QoR-15 test scores responses on a scale where 10 represents "always," and 0 means "never." The test has a maximum possible score of 150 and a minimum of 0. QoR-15 scores are classified into the following categories: excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121), and poor (QoR-15 < 90).

CONTACTS AND LOCATIONS:
Locations (1):
- VKV American Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All shared data will be de-identified to protect participant confidentiality, and access will be granted only to researchers who meet the necessary criteria and ethical standards for data use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The start date for IPD sharing will be after the completion of the study and the publication of the main study results, approximately June 2025.
  End Date for IPD Sharing: IPD will be available for sharing for a period of 5 years following the publication of the study results, until June 2030.
  During this period, researchers who meet the criteria for access will be able to request the de-identified data for secondary analyses.

REFERENCES:
- [Background] Çuhadaroğlu, F. (1986). Adolesanlarda benlik saygısı. Yayınlanmamış uzmanlık tezi. Hacettepe Üniversitesi.
- [Result] Miller MD, Ferris DG. Measurement of subjective phenomena in primary care research: the Visual Analogue Scale. Fam Pract Res J. 1993 Mar;13(1):15-24. PMID 8484338
- [Result] Kara U, Simsek F, Kamburoglu H, Ozhan MO, Alakus U, Ince ME, Eksert S, Ozkan G, Eskin MB, Senkal S. Linguistic validation of a widely used recovery score: quality of recovery-15 (QoR-15). Turk J Med Sci. 2022 Apr;52(2):427-435. doi: 10.55730/1300-0144.5330. Epub 2022 Apr 14. PMID 36161615
- [Result] Karakas Ugurlu G, Ugurlu M, Erten S, Can SS, Ulusoy Kaymak S, Caykoylu A. Effect of familial Mediterranean fever on sexual and reproductive health in women. Turk J Med Sci. 2017 Apr 18;47(2):463-469. doi: 10.3906/sag-1602-88. PMID 28425232
- [Result] Aydemir, O. J. T. P. D. (1997). Hastane anksiyete ve depresyon olcegi Turkce formunun gecerlilik ve guvenilirligi. Turk Psikiyatri Derg., 8, 187-280.
- [Result] Atak, H. (2013). On-Maddeli Kişilik Ölçeği'nin Türk Kültürü'ne Uyarlanması. Archives of Neuropsychiatry/Nöropsikiyatri Arşivi, 50(4).
- [Result] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Result] Schreiber KL, Zinboonyahgoon N, Xu X, Spivey T, King T, Dominici L, Partridge A, Golshan M, Strichartz G, Edwards RR. Preoperative Psychosocial and Psychophysical Phenotypes as Predictors of Acute Pain Outcomes After Breast Surgery. J Pain. 2019 May;20(5):540-556. doi: 10.1016/j.jpain.2018.11.004. Epub 2018 Nov 23. PMID 30476655
- [Result] Kam O, Na S, La Sala M, Tejeda CI, Koola MM. The Psychological Benefits of Cosmetic Surgery. J Nerv Ment Dis. 2022 Jul 1;210(7):479-485. doi: 10.1097/NMD.0000000000001477. PMID 35766540
- [Result] Honigman RJ, Phillips KA, Castle DJ. A review of psychosocial outcomes for patients seeking cosmetic surgery. Plast Reconstr Surg. 2004 Apr 1;113(4):1229-37. doi: 10.1097/01.prs.0000110214.88868.ca. PMID 15083026
- [Result] Kulkarni AR, Pusic AL, Hamill JB, Kim HM, Qi J, Wilkins EG, Roth RS. Factors Associated with Acute Postoperative Pain Following Breast Reconstruction. JPRAS Open. 2017 Mar;11:1-13. doi: 10.1016/j.jpra.2016.08.005. Epub 2016 Sep 15. PMID 28713853
- [Result] Bradshaw P, Hariharan S, Chen D. Does preoperative psychological status of patients affect postoperative pain? A prospective study from the Caribbean. Br J Pain. 2016 May;10(2):108-15. doi: 10.1177/2049463716635680. Epub 2016 Mar 2. PMID 27551421
- [Result] Aglio LS, Mezzalira E, Mendez-Pino L, Corey SM, Fields KG, Abbakar R, Baez LA, Kelly-Aglio NJ, Vetter T, Jamison RN, Edwards RR. Surgical Prehabilitation: Strategies and Psychological Intervention to Reduce Postoperative Pain and Opioid Use. Anesth Analg. 2022 May 1;134(5):1106-1111. doi: 10.1213/ANE.0000000000005963. No abstract available. PMID 35427271
- [Result] Williams ACC, Craig KD. Updating the definition of pain. Pain. 2016 Nov;157(11):2420-2423. doi: 10.1097/j.pain.0000000000000613. No abstract available. PMID 27200490